CLINICAL TRIAL: NCT02143414
Title: A Phase 2 Study of Blinatumomab and POMP (Prednisone, Vincristine, Methotrexate, 6-Mercaptopurine) for Patients >/= 65 Years of Age With Newly Diagnosed Philadelphia-Chromosome Negative (Ph-) Acute Lymphoblastic Leukemia (ALL) and of Dasatinib, Prednisone and Blinatumomab for Patients >/= 65 Years of Age With Newly Diagnosed Philadelphia-Chromosome Positive (Ph+) ALL, Relapsed/Refractory Ph+ ALL, and Philadelphia-Chromosome-Like Signature (Ph-Like) ALL (Newly Diagnosed or Relapsed/Refractory) With Known or Presumed Activating Dasatinib-Sensitive Mutations or Kinase Fusions (DSMKF)
Brief Title: Blinatumomab and Combination Chemotherapy or Dasatinib, Prednisone, and Blinatumomab in Treating Older Patients With Acute Lymphoblastic Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-01047; NCI-2014-01047 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); SWOG-S1318; S1318 (Other: SWOG); S1318 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2014-05-19; First posted 2014-05-21 (Estimated); Results first posted 2023-01-25 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Acute Lymphoblastic Leukemia; B Acute Lymphoblastic Leukemia; B Acute Lymphoblastic Leukemia With t(9;22)(q34.1;q11.2); BCR-ABL1; Recurrent Acute Lymphoblastic Leukemia; Refractory Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma | interventions — Biopsy; Specimen Handling; blinatumomab; N,N-dicyclohexyl-isoborneol-10-sulfonamide; Dasatinib; Spinal Puncture; Magnetic Resonance Spectroscopy; Mercaptopurine; azathiopurine; Methotrexate; merphos; Prednisone; deltacortene; prednylidene; Vincristine; X-Rays; Phantoms, Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort I (blinatumomab, POMP) (Experimental): See Detailed Description
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Biological: Blinatumomab; Procedure: Bone Marrow Aspiration and Biopsy; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Lumbar Puncture; Procedure: Magnetic Resonance Imaging; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Methotrexate Sodium; Drug: Prednisone; Drug: Vincristine; Drug: Vincristine Sulfate; Procedure: X-Ray Imaging
- Cohort II (dasatinib, prednisone, blinatumomab) (Experimental): See Detailed Description
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Biological: Blinatumomab; Procedure: Bone Marrow Aspiration and Biopsy; Procedure: Computed Tomography; Drug: Dasatinib; Procedure: Echocardiography Test; Procedure: Lumbar Puncture; Procedure: Magnetic Resonance Imaging; Drug: Prednisone; Procedure: X-Ray Imaging

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo a biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo a blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Biological: Blinatumomab — Given IV
  Other Names: AMG 103; AMG-103; AMG103; Anti-CD19 x Anti-CD3 Bispecific Monoclonal Antibody; Anti-CD19/Anti-CD3 Recombinant Bispecific Monoclonal Antibody MT103; Blincyto; MEDI 538; MEDI-538; MEDI538; MT 103; MT-103; MT103
Procedure: Bone Marrow Aspiration and Biopsy — Undergo a bone marrow aspiration and biopsy
Procedure: Computed Tomography — Undergo a CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Dasatinib — Given PO
  Other Names: BMS 354825; BMS-354825; BMS354825; Dasatinib Hydrate; Dasatinib Monohydrate; Sprycel
  Arms: Cohort II (dasatinib, prednisone, blinatumomab)
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Procedure: Lumbar Puncture — Undergo a lumbar puncture
  Other Names: LP; Spinal Tap
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Mercaptopurine — Given PO
  Other Names: 3H-Purine-6-thiol; 6 MP; 6 Thiohypoxanthine; 6 Thiopurine; 6-Mercaptopurine; 6-Mercaptopurine Monohydrate; 6-MP; 6-Purinethiol; 6-Thiopurine; 6-Thioxopurine; 6H-Purine-6-thione, 1,7-dihydro- (9CI); 7-Mercapto-1,3,4,6-tetrazaindene; Alti-Mercaptopurine; Azathiopurine; Bw 57-323H; Flocofil; Ismipur; Leukerin; Leupurin; Mercaleukim; Mercaleukin; Mercaptina; Mercaptopurinum; Mercapurin; Mern; NCI-C04886; Puri-Nethol; Purimethol; Purine, 6-mercapto-; Purine-6-thiol (8CI); Purine-6-thiol, monohydrate; Purinethiol; Purinethol; U-4748; WR-2785
  Arms: Cohort I (blinatumomab, POMP)
Drug: Methotrexate — Given PO
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Jylamvo; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
  Arms: Cohort I (blinatumomab, POMP)
Drug: Methotrexate Sodium — Given PO
  Other Names: Sodium Methotrexate; Trexall; Xatmep
  Arms: Cohort I (blinatumomab, POMP)
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Drug: Vincristine — Given IV
  Other Names: LCR; Leurocristine; VCR; Vincrystine
  Arms: Cohort I (blinatumomab, POMP)
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate
  Arms: Cohort I (blinatumomab, POMP)
Procedure: X-Ray Imaging — Undergo an x-ray
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Plain film radiographs; Radiographic Imaging; Radiographic imaging procedure (procedure); Radiography; RG; Static X-Ray; X-Ray

SUMMARY:
This phase II trial studies the side effects and how well blinatumomab and combination chemotherapy or dasatinib, prednisone, and blinatumomab work in treating older patients with acute lymphoblastic leukemia. Immunotherapy with monoclonal antibodies, such as blinatumomab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Chemotherapy drugs, such as prednisone, vincristine sulfate, methotrexate, and mercaptopurine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Dasatinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving blinatumomab with combination chemotherapy or dasatinib and prednisone may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the 3-year survival rate in elderly patients with newly diagnosed Philadelphia (Ph)-negative acute lymphoblastic leukemia (ALL) treated with blinatumomab followed by POMP (prednisone, vincristine sulfate, methotrexate, and mercaptopurine) maintenance.

II. To evaluate in a preliminary manner (feasibility study) the safety of dasatinib-steroid based induction followed by blinatumomab treatment in combination with dasatinib followed by dasatinib-based maintenance in patients with newly diagnosed Ph-positive ALL, relapsed/refractory Ph-positive ALL, and Ph-like dasatinib-sensitive mutations or kinase fusions (DSMKF) ALL (newly-diagnosed relapsed or refractory).

SECONDARY OBJECTIVES:

I. To evaluate toxicities in these patient populations treated with these regimens.

II. To estimate the rates of complete response (CR), complete remission with incomplete count recovery (CRi) and disease-free survival in Ph-negative patients.

III. To estimate disease-free and overall survival in Ph-positive ALL and Ph-like DSMKF ALL.

IV. To estimate in each cohort the rate of minimal residual disease (MRD) negativity, and the time to achieve MRD negativity (exploratory analysis).

V. To determine whether anti-idiotype antibodies directed against blinatumomab develop with blinatumomab treatment in this study.

ADDITIONAL TRANSLATIONAL MEDICINE OBJECTIVES:

I. To estimate the incidence of the Ph-like signature in elderly patients (>= 65 years of age) with newly diagnosed Philadelphia-chromosome negative ALL.

II. To estimate the incidence of the various tyrosine-kinase fusions, making up the Ph-like signature in elderly patients with newly diagnosed Philadelphia-chromosome negative ALL.

III. To evaluate outcomes (event free survival [EFS] and overall survival [OS]) in patients with the Ph-like signature versus those without the Ph-like signature in Ph-negative ALL.

IV. To describe via single cell transcriptomics the clonal diversity in gene expression of participants on the trial.

V. To describe the methylation status of the overall genome as well as key driver genes of all participants in the trial.

OUTLINE: Patients are assigned to 1 of 2 treatment cohorts according to Philadelphia chromosome status.

COHORT I (PHILADELPHIA CHROMOSOME NEGATIVE PATIENTS):

INDUCTION: Patients receive blinatumomab intravenously (IV) continuously over 24 hours on days 1-28 in the absence of disease progression or unacceptable toxicity. Patients undergo an x-ray and echocardiography (ECHO) during screening and a computed tomography (CT) scan and/or magnetic resonance imaging (MRI) as well as blood sample collection and bone marrow aspiration and biopsy throughout the trial. Patients undergo a lumbar puncture during screening and on study. Patients may also undergo a biopsy during screening. (Closed to accrual 06/29/17)

RE-INDUCTION: Patients not achieving CR or CRi after Induction, receive blinatumomab IV continuously over 24 hours on days 1-28 in the absence of disease progression or unacceptable toxicity. Patients undergo an x-ray and ECHO during screening and a CT scan and/or MRI as well as blood sample collection and bone marrow aspiration and biopsy throughout the trial. Patients undergo a lumbar puncture during screening and on study. Patients may also undergo a biopsy during screening.

POST-REMISSION: Patients receive blinatumomab IV continuously over 24 hours on days 1-28. Treatment repeats every 42 days for 3 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo a CT scan and/or MRI on study and during follow-up. Patients also undergo blood sample collection, lumbar puncture, and bone marrow aspiration and biopsy on study.

MAINTENANCE: Patients receive prednisone orally (PO) on days 1-5, vincristine sulfate IV on day 1, mercaptopurine PO on days 1-28, and methotrexate PO on days 1, 8, 15, and 22. Treatment repeats every 28 days for 18 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo a CT scan and/or MRI on study and during follow-up. Patients also undergo a lumbar puncture and bone marrow aspiration and biopsy on study.

COHORT II (PHILADELPHIA CHROMOSOME POSITIVE PATIENTS):

INDUCTION: Patients receive dasatinib PO on days 1-84 and prednisone PO on days 1-24 with tapering on days 25-32 in the absence of disease progression or unacceptable toxicity. Patients undergo an x-ray and ECHO during screening and a CT scan and/or MRI throughout the trial. Patients undergo a lumbar puncture and bone marrow aspiration and biopsy during screening and on study. Patients may also undergo a biopsy during screening.

RE-INDUCTION: Patients receive blinatumomab IV continuously over 24 hours on days 1-28. Treatment repeats every 42 days for 2 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo a CT scan and/or MRI on study and during follow-up. Patients also undergo blood sample collection, a lumbar puncture, and bone marrow aspiration and biopsy on study.

POST-REMISSION: Patients receive blinatumomab IV continuously over 24 hours on days 1-28 and dasatinib PO on days 1-42. Treatment repeats every 42 days for 3 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo a CT scan and/or MRI on study and during follow-up. Patients also undergo blood sample collection, lumbar puncture, and bone marrow aspiration and biopsy on study.

MAINTENANCE: Patients receive dasatinib PO on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also receive prednisone PO on days 1-5. Treatment repeats every 28 days for 18 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo a CT scan and/or MRI as well as a lumbar puncture and bone marrow aspiration and biopsy on study.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 2 years, and then annually until 10 years from initial registration.

ELIGIBILITY:
Inclusion Criteria:

* Registration Step 1 - Induction/Re-Induction:
* Patients must have a new morphologic diagnosis of precursor B cell acute lymphoblastic leukemia (ALL) (non T cell) based on World Health Organization (WHO) criteria; patients with Burkitt's (L3) are excluded; patients with Ph-positive or Ph-like ALL with dasatinib-sensitive mutations or kinase fusions may have relapsed or refractory diagnoses

  * NOTE: Relapsed/refractory Ph-positive patients or Ph-like patients with dasatinib-sensitive mutations or kinase fusions who have previous exposure to either dasatinib or another 2nd or 3rd generation tyrosine kinase inhibitor (TKI) will begin protocol therapy with Cohort 2: re-induction cycle 1
* Patients must have a diagnosis of Philadelphia chromosome negative ALL or Ph chromosome positive ALL by cytogenetics, fluorescence in situ hybridization (FISH) or polymerase chain reaction (PCR); patients will be registered to receive treatment in either Cohort 1 (Ph-) or Cohort 2 (Ph+ or Ph-like DSMKF) based on these results; diagnostic specimens must be submitted to the site's local Clinical Laboratory Improvement Amendments (CLIA)-approved cytogenetics laboratory and results of tests (cytogenetics, FISH or PCR) must confirm Ph status prior to registration; if not already known, breakpoint cluster region- abelson murine leukemia viral oncogene homolog 1 (BCR-ABL) status (p190 or p210) must be evaluated in Ph-positive patients by PCR

  * For Cohort 2, Ph-like testing is not required specifically for this study; however, to be registered to Cohort 2 under the Ph-like DSMKF criterion, the patient must have a known or presumed activating Ph-like signature and dasatinib-sensitive mutation or kinase fusion, such as: ABL1, ABL2, colony stimulating factor 1 receptor (CSF1R), platelet derived growth factor receptor beta (PDGFRB), platelet derived growth factor receptor alpha (PDGFRA), or fibroblast growth factor receptor (FGFR)s that was otherwise identified as part of normal standard of care; prior to registering any patients with a known or presumed activating Ph-like signature and dasatinib-sensitive mutations or kinase fusions (DSMKF) treating physicians must confirm eligibility with the study chairs via email; the study chairs must respond via email with confirmation of patient eligibility prior to patient registration
* All newly diagnosed patients must have evidence of ALL in their marrow or peripheral blood with at least 20% lymphoblasts present in blood or bone marrow collected within 28 days prior to registration; all relapsed/refractory patients (Cohort 2) must have at least 5% lymphoblasts present in blood or bone marrow collected within 28 days prior to registration; for relapsed/refractory patients, pathology and cytogenetics reports (both from time of original diagnosis) must be submitted at time of registration; if a bone marrow aspirate cannot be obtained despite an attempt (dry tap), appropriate immunohistochemistry (IHC) testing, including cluster of differentiation (CD)19, must be performed on the bone marrow biopsy to determine lineage; for ALL in marrow or peripheral blood, immunophenotyping of the blood or marrow lymphoblasts must be performed to determine lineage (B cell, T cell or mixed B/T cell); appropriate marker studies including CD19 (B cell), must be performed; co-expression of myeloid antigens (CD13 and CD33) will not exclude patients; if possible, the lineage specific markers (myeloid cells) should be determined; the blood/bone marrow sample for these assays must be obtained within 28 days prior to registration; patients with only extramedullary disease in the absence of bone marrow or blood involvement are not eligible
* Patient must not have a history or presence of clinically relevant central nervous system (CNS) pathology such as epilepsy, seizure, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, psychosis, active ALL in the CNS confirmed by cerebrospinal fluid (CSF) analysis, or other significant CNS abnormalities
* Patients must have a lumbar puncture to determine CNS involvement of ALL within 14 days prior to registration; patients with CNS3 are excluded from the trial; patients with CNS1 or CNS2 will be eligible, but will be monitored for CNS involvement; note that intrathecal methotrexate administered during the pre-study lumbar puncture may count as the first dose of intrathecal therapy required as part of the study
* Cohort I, Ph-negative Patients Only: Patients must not have received any prior chemotherapy, radiation therapy, or other therapy for the treatment of ALL (other than those noted below) and must not be receiving any immunosuppressive therapy; patients may not have received any prior investigational therapy within 28 days prior to registration; patients must not have received any monoclonal antibody therapy within 42 days of registration; patients may have received the following within any time prior to registration: low dose chemotherapy-including: cyclophosphamide 1 g/m^2, oral 6-mercaptopurine, or oral methotrexate (other low dose chemotherapy may be allowable, however any other options not listed here should be confirmed with the study chairs), TKI therapy, steroids, hydroxyurea, leukapheresis, intrathecal chemotherapy or vincristine
* Cohort I, Ph-negative Patients Only: In the event that the patient's bone marrow blast count is >= 50% blasts, patients may be registered but should receive steroids for 3-5 days in order to reduce tumor burden prior to blinatumomab administration, as follows

  * Prephase treatment with dexamethasone (10-20 mg/m^2) for 3-5 days is required for patients with bone marrow blasts >= 50%, peripheral blood blasts 15,000/uL or higher, or elevated lactate dehydrogenase (LDH) suggesting rapidly progressive disease per investigator opinion

    * Pre-treatment should conclude at least 24 hours prior to the first dose of blinatumomab (although additional dexamethasone is automatically given as a pre-med prior to the first dose); at the time of first infusion of blinatumomab, the absolute peripheral blast count should be < 25,000/uL
    * Note: For the purposes of the study, day 1 of the cycle will be the first day of blinatumomab administration
* Cohort I, Ph-negative Patients Only: It is preferred, but not required, that corticosteroids and hydroxyurea should start only after all diagnostic samples have been obtained; however, if the patient was previously on corticosteroids and/or hydroxyurea, this is allowable provided that the patient still has measurable disease at time of the bone marrow aspirate

  * Corticosteroids and/or hydroxyurea, as well as any of the other therapies mentioned (with the exception of IV cyclophosphamide), may continue to be administered, at physician discretion, until 1 day prior to blinatumomab administration
  * IV cyclophosphamide must be discontinued at least 7 days prior to blinatumomab administration
* Cohort 2, Ph-positive and Ph-like DSMKF Patients Only: Patients must NOT have received a prior autologous or allogeneic hematopoietic stem cell transplant at any time. Patients must NOT have received any chemotherapy, investigational agents, or undergone major surgery within 14 days prior to registration, with the following exceptions:

  * Monoclonal antibodies must not have been received for 1 week prior to registration
  * Chimeric antigen receptor (CAR) T-cells must not have been received for 28 days prior to registration
  * Steroids, hydroxyurea, vincristine, 6-mercaptopurine, methotrexate, thioguanine and intrathecal chemotherapy are permitted within any timeframe prior to registration; Food and Drug Administration (FDA)-approved TKIs may also be administered until 1 day prior to start of study therapy (C1, D1); IV cyclophosphamide may be administered at doses of 1 g/m^2 or less until up to 7 days prior to registration
* Patients must be >= 65 years of age; for patients 65-69 years of age, patient must be deemed not suitable for standard intensive induction chemotherapy at the discretion of the local investigator, or must have refused standard intensive chemotherapy
* Cohort I, Ph-negative Patients Only: Patients must not be candidates for allogeneic hematopoietic stem cell transplant; NOTE: Subjects up to age 70 years who are considered fit for allogeneic hematopoietic stem cell transplant, should be considered for enrollment on E1910, in order to avoid competing with that study; if a patient is considered unfit for intensive chemotherapy at the time of initial diagnosis, but subsequently achieves a complete remission (CR), then it will be left to the treating physician's discretion to consider hematopoietic stem cell transplant (HSCT)
* Cohort I, Ph-negative Patients Only: Patients must have complete history and physical examination within 28 days prior to registration
* Cohort I, Ph-negative Patients Only: Patients must have a Zubrod performance status of 0-2
* Cohort I, Ph-negative Patients Only: Patients must have serum creatinine =< 1.5 mg/dl within 14 days prior to registration
* Cohort I, Ph-negative Patients Only: Patients must have aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3.0 x institutional upper limit of normal (IULN) within 14 days prior to registration
* Cohort I, Ph-negative Patients Only: Patients must have total bilirubin =< 2.0 x IULN within 14 days prior to registration
* Cohort I, Ph-negative Patients Only: Patients must have alkaline phosphatase =< 2.5 x IULN within 14 days prior to registration
* Cohort I, Ph-negative Patients Only: Patients must not have systemic fungal, bacterial, viral or other infection that is not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment)
* Cohort I, Ph-negative Patients Only: Patients must not have Common Terminology Criteria for Adverse Events (CTCAE) >= grade 2 neuropathy (cranial, motor or sensory) within 14 days prior to registration
* Cohort I, Ph-negative Patients Only: Patients known to be positive for HIV (the human immunodeficiency virus) may be eligible, providing they meet the following additional criteria within 28 days prior to registration:

  * No history of acquired immune deficiency syndrome (AIDS)-defining conditions
  * CD4 cells > 350 cells/mm^3
  * If on antiretroviral agents, must not include zidovudine or stavudine
  * Viral load =< 50 copies HIV messenger ribonucleic acid (mRNA)/mm^3 if on combination antiretroviral therapy (cART) or =< 25,000 copies HIV mRNA/mm^3 if not on cART
  * Highly active antiretroviral therapy (HAART) regimens are acceptable providing they have only weak P450A4 interactions
* Cohort I, Ph-negative Patients Only: Patients must not have any known autoimmune disease
* Cohort I, Ph-negative Patients Only: Patients must not have testicular involvement; if clinical or ultrasound findings are equivocal, biopsy must be performed; all tests for establishing testicular involvement must be completed within 14 days prior to registration
* Cohort I, Ph-negative Patients Only: Patients with evidence of extramedullary disease at diagnosis will have computed tomography (CT) scan or magnetic resonance imaging (MRI) of the chest, abdomen and pelvis to obtain baseline values within 28 days prior to registration
* Cohort I, Ph-negative Patients Only: No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for five years
* Cohort I, Ph-negative Patients Only: Patients must have the following tests within 28 days prior to registration to obtain baseline measurements:

  * Prothrombin time (PT)/partial thromboplastin time (PTT)/international normalized ratio (INR)/fibrinogen (all patients)
  * Cohort 1, Ph- Patients Only: Neurologic assessment
* Cohort 2, Ph+ and Ph-like DSMKF Patients Only: Patients must not have active pericardial effusion, ascites or pleural effusion of any grade based on chest x-ray and echocardiogram within 28 days prior to registration; exception: if the effusion is suspected to be related to the leukemia, the patient may have pericardial effusion =< grade 2 or pleural effusion =< grade 1
* Cohort 2, Ph+ and Ph-like DSMKF Patients Only: Patients must have ejection fraction >= 45% based on echocardiogram performed within 28 days prior to registration
* Cohort 2, Ph+ and Ph-like DSMKF Patients Only: Patients must have QTcF (by Fridericia calculation) < 480/msec based on electrocardiogram (EKG) performed within 28 days prior to registration
* Cohort 2, Ph+ and Ph-like DSMKF Patients Only: Patients must not be receiving any proton pump inhibitors at the time of registration
* Pretreatment cytogenetics must be performed on all patients; collection of pretreatment specimens must be completed within 28 days prior to registration to S1318; specimens must be submitted to the site's preferred CLIA-approved cytogenetics laboratory; BCR-ABL status must be verified in Ph-positive patients by FISH, cytogenetics, and/or PCR prior to enrollment; if a patient is Ph-positive, PCR for both p190 and p210 must be sent
* Patients must be offered participation in specimen submission for future research; with patient's consent, specimens must be submitted as outlined
* Cohort 1, Ph-negative Patients Only: Patients must have specimens submitted for blinatumomab immunogenicity assessment; collection of pretreatment specimens must be completed within 28 days prior to registration to S1318; specimens must be submitted to LabConnect
* Cohort 2, Ph-positive and Ph-like DSMKF Patients Only: Patients must agree to have specimens submitted for blinatumomab immunogenicity testing if subsequently moved to a blinatumomab containing treatment regimen on protocol
* Patients or their legally authorized representative must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system
* Registration Step 2 - Post-Remission Therapy:
* Cohort 1, Ph-negative Patients Only: Patients must have achieved CR or CRi within 2 cycles of induction/re-induction with blinatumomab

  * NOTE: day 1 of post-remission = day 43 of the preceding cycle (+/- 3 days)
* Cohort 2, Ph-positive and Ph-like DSMKF Patients Only: Newly diagnosed Ph+, newly-diagnosed Ph-like DSMKF, and relapsed/refractory Ph+ patients without prior dasatinib or other 2nd or 3rd generation TKI therapy, must have achieved CR or CRi within 1 cycle of induction with dasatinib/prednisone, or within 2 cycles of re-induction with blinatumomab; relapsed/refractory Ph+ or Ph-like DSMKF patients with prior dasatinib or other 2nd or 3rd generation TKI therapy must have achieved CR or CRi within 2 cycles of re-induction therapy with blinatumomab

  * NOTE: day 1 of post-remission = day 85 of the preceding induction cycle (+/- 3 days), or day 43 of the preceding re-induction cycle (+/- 3 days) as applicable
* Serum creatinine =< 1.5 mg/dl within 14 days prior to registration
* AST and ALT =< 3.0 x institutional upper limit of normal (IULN) within 14 days prior to registration
* Total bilirubin =< 2.0 x IULN within 14 days prior to registration
* Absolute neutrophil count (ANC) >= 750/mcL within 28 days prior to registration
* Platelets >= 50,000/mcL within 28 days prior to registration
* Patients must be registered to Step 2 within 28 days after count recovery; (Note: there is no maximum allotted time period for count recovery, providing patient remains in CR or CRi)
* All non-hematologic treatment related toxicities that are deemed clinically significant by the treating investigator must have resolved to =< grade 2
* Registration Step 3 - Maintenance: Patients must have documented CR or CRi within 28 days prior to registration; note that bone marrow examination is only required if there are clinical signs/symptoms of progression; if progression is a concern due to the length of the time for count recovery, a bone marrow examination is recommended
* Registration Step 3 - Maintenance: Patients must have serum creatinine =< 1.5 mg/dl within 14 days prior to registration
* Registration Step 3 - Maintenance: Patients must have AST and ALT =< 3.0 x institutional upper limit of normal (IULN) within 14 days prior to registration
* Registration Step 3 - Maintenance: Patients must have total bilirubin < 2.0 x institutional upper limit of normal (IULN) within 14 days prior to registration
* Registration Step 3 - Maintenance: Patients must have adequate marrow function as evidenced by ANC >= 750/mcL within 28 days prior to registration
* Registration Step 3 - Maintenance: Patients must have adequate marrow function as evidenced by platelets >= 75,000/mcL within 28 days prior to registration
* Registration Step 3 - Maintenance: All non-hematologic treatment related toxicities that are deemed clinically significant by the treating investigator must have resolved to =< grade 2

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 53 (Actual)
Dates: Start 2015-06-30 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2026-06-24 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Anjali S Advani, Principal Investigator — SWOG Cancer Research Network
Locations (196):
- United States (196):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - John L McClellan Memorial Veterans Hospital, Little Rock, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Keck Medical Center of USC Pasadena, Pasadena, California
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Orlando Health Cancer Institute, Orlando, Florida
  - Northside Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Rush-Copley Medical Center, Aurora, Illinois
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Reid Health, Richmond, Indiana
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Hickman Cancer Center, Adrian, Michigan
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Corewell Health Farmington Hills Hospital, Farmington Hills, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - William Beaumont Hospital-Grosse Pointe, Grosse Pointe, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - University of Rochester, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - ECU Health Oncology Kenansville, Kenansville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - ECU Health Oncology Richlands, Richlands, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Miami Valley Hospital South, Centerville, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Baylor University Medical Center, Dallas, Texas
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Advani AS, Moseley A, O'Dwyer KM, Wood BL, Park J, Wieduwilt M, Jeyakumar D, Yaghmour G, Atallah EL, Gerds AT, O'Brien SM, Liesveld JL, Othus M, Litzow M, Stone RM, Sharon E, Erba HP. Dasatinib/prednisone induction followed by blinatumomab/dasatinib in Ph+ acute lymphoblastic leukemia. Blood Adv. 2023 Apr 11;7(7):1279-1285. doi: 10.1182/bloodadvances.2022008216. PMID 36322825

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 57 total participants registered to the study; 31 in Cohort I and 26 in Cohort II. Four participants, two from each cohort, were deemed ineligible at the start of the study and never received protocol treatment. This left 53 eligible participants; 29 in Cohort II and 24 in Cohort II.
Groups:
- Cohort I (Ph-): INDUCTION: Patients receive blinatumomab IV continuously over 24 hours on days 1-28 in the absence of disease progression or unacceptable toxicity.
  RE-INDUCTION: Patients not achieving CR or CRi after Induction, receive blinatumomab IV continuously over 24 hours on days 1-28 in the absence of disease progression or unacceptable toxicity.
  POST-REMISSION: Patients receive blinatumomab IV continuously over 24 hours on days 1-28. Treatment repeats every 42 days for 3 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Patients receive prednisone PO on days 1-5, vincristine sulfate IV on day 1, mercaptopurine PO on days 1-28, and methotrexate PO on days 1, 8, 15, and 22. Treatment repeats every 28 days for 18 cycles in the absence of disease progression or unacceptable toxicity. (Closed to accrual 06/29/17)
  Blinatumomab: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Mercaptopurine: Given PO
  Methotrexate: Given PO
  Methotrexate Sodium: Given PO
  Prednisone: Given PO
  Vincristine: Given IV
  Vincristine Sulfate: Given IV
- Cohort II (Ph+/Ph-like): INDUCTION: Patients receive dasatinib PO BID on days 1-84 and prednisone PO on days 1-24 with tapering on days 25-32 in the absence of disease progression or unacceptable toxicity.
  RE-INDUCTION: Patients receive blinatumomab IV continuously over 24 hours on days 1-28. Treatment repeats every 42 days for 2 cycles in the absence of disease progression or unacceptable toxicity.
  POST-REMISSION: Patients receive blinatumomab IV continuously over 24 hours on days 1-28 and dasatinib PO QD on days 1-42. Treatment repeats every 42 days for 3 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Patients receive dasatinib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also receive prednisone PO on days 1-5. Treatment repeats every 28 days for 18 cycles in the absence of disease progression or unacceptable toxicity.
  Blinatumomab: Given IV
  Dasatinib: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Prednisone: Given PO
Period: Induction
Arm/Group | Cohort I (Ph-) | Cohort II (Ph+/Ph-like)
Started | 29 | 24
Completed Induction | 24 | 19
Completed | 19 | 18
Not Completed | 10 | 6
Not completed — Adverse Event | 1 | 2
Not completed — Death | 1 | 2
Not completed — Patient refusal | 1 | 1
Not completed — Refractory | 1 | 0
Not completed — Began alternative treatment | 1 | 0
Not completed — Ineligible for postremission | 5 | 1
Period: Post-remission
Arm/Group | Cohort I (Ph-) | Cohort II (Ph+/Ph-like)
Started | 19 | 18
Completed | 14 | 16
Not Completed | 5 | 2
Not completed — Adverse Event | 0 | 2
Not completed — Disease progression/relapse | 5 | 0
Period: Maintenance
Arm/Group | Cohort I (Ph-) | Cohort II (Ph+/Ph-like)
Started | 14 | 16
Completed | 4 | 0
Not Completed | 10 | 16
Not completed — Adverse Event | 4 | 6
Not completed — Disease progression/relapse | 3 | 2
Not completed — Patient refusal | 2 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Death | 0 | 1
Not completed — On protocol treatment | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort I (Ph-) | Cohort II (Ph+/Ph-like) | Total
Number analyzed (Participants) | 29 | 24 | 53
Age, Continuous [Median (Full Range); unit: years] | 75.4 [66.3 to 84.0] | 73.5 [65.0 to 87.2] | 74.7 [65.0 to 87.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 16 | 23
  Male | 22 | 8 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 27 | 18 | 45
  Unknown or Not Reported | 0 | 3 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 28 | 18 | 46
  Black | 0 | 1 | 1
  Asian | 1 | 2 | 3
  Unknown | 0 | 3 | 3
Baseline WBC [Median (Full Range); unit: 10^3 cells/uL] — Baseline white blood cell (WBC) count
  10^3 cells/uL | 3.0 [0.3 to 520.8] | 7.5 [1.3 to 123.3] | 5.1 [0.3 to 520.8]
Baseline Marrow Blasts [Median (Full Range); unit: percentage] | 87 [30 to 100] | 88.5 [30 to 100] | 88.4 [30 to 100]

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival Rate (Cohort I)
Description: To evaluate the 3-year overall survival rate in elderly participants with newly diagnosed Ph-negative ALL treated with blinatumomab followed by POMP maintenance. Overall
Time Frame: From the day of registration on study until death from any cause, assessed at 3 years
Population: Only participants in Cohort I were evaluated
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort I (Ph-)
Number analyzed (Participants) | 29
percentage of participants | 34 [18 to 54]

2. Primary Outcome: Incidence of Dose-limiting Toxicity (Cohort II)
Description: Defined as any grade 4 or higher treatment-related, non-hematologic toxicity in the first cycle of post-remission therapy (blinatumomab/dasatinib) graded by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Only participants with Ph-positive ALL or Ph-like DSMKF ALL were evaluated.
Time Frame: Up to day 42 of post-remission therapy
Population: Only participants in Cohort II that registered to post-remission were analyzed for dose-limiting toxicities.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort II (Ph+/Ph-like)
Number analyzed (Participants) | 18
Participants | 0

3. Secondary Outcome: Number of Participants With Grade 3 Through 5 Adverse Events That Are Related to Study Drugs
Description: Number of participants with Grade 3-5 adverse events that are possibly, probably or definitely related to study drug are reported by given type of adverse event. Adverse Events reported using CTCAE v 4.0, whereas Serious Adverse Events were reported with CTCAE v 5.0.
Time Frame: Duration of treatment and follow up until death or date of primary analysis (about 7.5 years)
Population: Eligible participants who received at least one dose of protocol treatment.
Measure: Number; unit: Participants
Groups:
- Induction: Cohort I (Ph-): INDUCTION: Patients receive blinatumomab IV continuously over 24 hours on days 1-28 in the absence of disease progression or unacceptable toxicity.
  RE-INDUCTION: Patients not achieving CR or CRi after Induction, receive blinatumomab IV continuously over 24 hours on days 1-28 in the absence of disease progression or unacceptable toxicity.
  Blinatumomab: Given IV
- Induction: Cohort II (Ph+/Ph-like): INDUCTION: Patients receive dasatinib PO BID on days 1-84 and prednisone PO on days 1-24 with tapering on days 25-32 in the absence of disease progression or unacceptable toxicity.
  RE-INDUCTION: Patients receive blinatumomab IV continuously over 24 hours on days 1-28. Treatment repeats every 42 days for 2 cycles in the absence of disease progression or unacceptable toxicity.
  Blinatumomab: Given IV
  Dasatinib: Given PO
  Prednisone: Given PO
- Post-remission: Cohort I (Ph-): POST-REMISSION: Patients receive blinatumomab IV continuously over 24 hours on days 1-28. Treatment repeats every 42 days for 3 cycles in the absence of disease progression or unacceptable toxicity.
  Blinatumomab: Given IV
- Post-remission: Cohort II (Ph+/Ph-like): POST-REMISSION: Patients receive blinatumomab IV continuously over 24 hours on days 1-28 and dasatinib PO QD on days 1-42. Treatment repeats every 42 days for 3 cycles in the absence of disease progression or unacceptable toxicity.
  Blinatumomab: Given IV
  Dasatinib: Given PO
- Maintenance: Cohort I (Ph-): MAINTENANCE: Patients receive prednisone PO on days 1-5, vincristine sulfate IV on day 1, mercaptopurine PO on days 1-28, and methotrexate PO on days 1, 8, 15, and 22. Treatment repeats every 28 days for 18 cycles in the absence of disease progression or unacceptable toxicity. (Closed to accrual 06/29/17)
  Mercaptopurine: Given PO
  Methotrexate: Given PO
  Methotrexate Sodium: Given PO
  Prednisone: Given PO
  Vincristine: Given IV
  Vincristine Sulfate: Given IV
- Maintenance: Cohort II (Ph+/Ph-like): MAINTENANCE: Patients receive dasatinib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also receive prednisone PO on days 1-5. Treatment repeats every 28 days for 18 cycles in the absence of disease progression or unacceptable toxicity.
  Dasatinib: Given PO
  Prednisone: Given PO
Arm/Group | Induction: Cohort I (Ph-) | Induction: Cohort II (Ph+/Ph-like) | Post-remission: Cohort I (Ph-) | Post-remission: Cohort II (Ph+/Ph-like) | Maintenance: Cohort I (Ph-) | Maintenance: Cohort II (Ph+/Ph-like)
Number analyzed (Participants) | 29 | 24 | 19 | 18 | 13 | 16
Participants
  Abdominal pain | 0 | 0 | 0 | 0 | 1 | 0
  Adult respiratory distress syndrome | 0 | 0 | 0 | 0 | 0 | 1
  Agitation | 0 | 0 | 0 | 1 | 0 | 0
  Alanine aminotransferase increased | 1 | 1 | 0 | 1 | 2 | 0
  Alkaline phosphatase increased | 0 | 0 | 0 | 0 | 0 | 1
  Anemia | 10 | 8 | 2 | 1 | 4 | 0
  Anorexia | 0 | 0 | 0 | 0 | 0 | 1
  Aspartate aminotransferase increased | 0 | 0 | 0 | 1 | 2 | 0
  Atrial flutter | 0 | 0 | 0 | 0 | 0 | 1
  Blood bilirubin increased | 0 | 0 | 0 | 0 | 2 | 0
  Cataract | 0 | 0 | 0 | 0 | 1 | 0
  Catheter related infection | 0 | 1 | 0 | 0 | 0 | 0
  Colitis | 0 | 0 | 0 | 0 | 1 | 1
  Confusion | 1 | 0 | 0 | 2 | 0 | 0
  Cytokine release syndrome | 1 | 0 | 0 | 0 | 0 | 0
  Dehydration | 0 | 1 | 0 | 0 | 0 | 1
  Diarrhea | 1 | 1 | 0 | 0 | 1 | 1
  Dizziness | 0 | 1 | 0 | 0 | 0 | 0
  Dysarthria | 1 | 0 | 0 | 0 | 0 | 0
  Dyspnea | 3 | 1 | 0 | 3 | 0 | 2
  Edema limbs | 0 | 2 | 0 | 0 | 0 | 0
  Encephalopathy | 0 | 0 | 0 | 1 | 0 | 0
  Fatigue | 1 | 0 | 1 | 0 | 3 | 0
  Febrile neutropenia | 3 | 1 | 0 | 0 | 2 | 0
  Fever | 1 | 0 | 0 | 0 | 0 | 0
  Gastrointestinal pain | 0 | 0 | 0 | 1 | 0 | 0
  General disorders and admin site conditions - Other | 0 | 1 | 0 | 0 | 0 | 1
  Generalized muscle weakness | 0 | 1 | 0 | 0 | 0 | 0
  Heart failure | 0 | 1 | 0 | 0 | 0 | 2
  Hematoma | 0 | 1 | 0 | 0 | 0 | 0
  Hyperglycemia | 4 | 1 | 1 | 2 | 1 | 0
  Hypertension | 3 | 0 | 1 | 2 | 1 | 4
  Hypoalbuminemia | 0 | 0 | 0 | 0 | 1 | 0
  Hypocalcemia | 1 | 0 | 0 | 1 | 0 | 0
  Hypokalemia | 0 | 1 | 1 | 0 | 0 | 0
  Hypophosphatemia | 1 | 0 | 0 | 0 | 1 | 0
  Hypotension | 1 | 1 | 0 | 0 | 0 | 0
  Hypoxia | 1 | 1 | 0 | 0 | 1 | 1
  Infections and infestations - Other, specify | 1 | 1 | 0 | 2 | 2 | 0
  Infusion related reaction | 1 | 0 | 0 | 0 | 0 | 0
  Lung infection | 2 | 2 | 0 | 0 | 1 | 1
  Lymphocyte count decreased | 8 | 6 | 2 | 6 | 4 | 0
  Metabolism and nutrition disorders - Other, specify | 0 | 0 | 0 | 0 | 0 | 1
  Mucositis oral | 0 | 0 | 0 | 0 | 1 | 0
  Nausea | 0 | 1 | 0 | 0 | 0 | 0
  Nervous system disorders - Other, specify | 1 | 0 | 0 | 0 | 0 | 0
  Neutrophil count decreased | 10 | 9 | 5 | 10 | 11 | 3
  Non-cardiac chest pain | 0 | 0 | 0 | 0 | 0 | 1
  Pericardial effusion | 0 | 0 | 0 | 1 | 0 | 1
  Platelet count decreased | 13 | 8 | 0 | 0 | 2 | 0
  Pleural effusion | 0 | 0 | 0 | 0 | 0 | 2
  Pneumonitis | 1 | 0 | 0 | 0 | 1 | 0
  Pulmonary hypertension | 0 | 0 | 0 | 0 | 0 | 1
  Rash maculo-papular | 0 | 1 | 0 | 0 | 0 | 0
  Respiratory failure | 1 | 0 | 0 | 0 | 1 | 0
  Sepsis | 0 | 1 | 0 | 0 | 2 | 0
  Soft tissue infection | 0 | 0 | 0 | 0 | 1 | 0
  Thrombotic thrombocytopenic purpura | 1 | 0 | 0 | 0 | 0 | 0
  Urinary tract infection | 0 | 1 | 0 | 0 | 0 | 0
  Vascular access complication | 0 | 0 | 0 | 0 | 1 | 0
  Weight loss | 0 | 0 | 0 | 0 | 0 | 1
  White blood cell decreased | 11 | 6 | 2 | 1 | 5 | 0

4. Secondary Outcome: Complete Response Rate (Cohort I)
Description: Complete response rate is measured by the number of participants achieving complete remission (CR) or complete remission with incomplete platelet recovery (CRi) rate. CR is defined as having <5% marrow aspirate blasts, ANC >1,000/mcL, platelets > 100,000/mcL, no blasts in peripheral blood, and C1 extramedullary disease status. CRi is the same as CR but platelet count may be <= 100,000/mcL and/or ANC <=1,000/mcL.
Time Frame: Participants are assessed after induction treatment and again after re-induction treatment, if re-induction treatment is received (i.e. up to 85 days after registration)
Population: Only participants in Cohort I were evaluated.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort I (Ph-)
Number analyzed (Participants) | 29
Participants
  CR or CRi | 19
  No CR or CRi | 10

5. Secondary Outcome: Disease-free Survival (Cohort II)
Description: An estimate of disease free survival in Ph-positive ALL and Ph-like DSMKF ALL (Cohort II). Disease free survival is measured by the number of years between the date the patient first achieves complete remission (CR) or complete remission with incomplete platelet recovery (CRi) until relapse from CR/CRi or death from any cause. CR is defined as having <5% marrow aspirate blasts, ANC >1,000/mcL, platelets > 100,000/mcL, no blasts in peripheral blood, and C1 extramedullary disease status. CRi is the same as CR but platelet count may be <= 100,000/mcL and/or ANC <=1,000/mcL.
Time Frame: Duration of treatment and follow up until death or date of primary analysis (about 7.5 years)
Population: Only participants in Cohort II that achieved complete remission were analyzable.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Cohort II (Ph+/Ph-like)
Number analyzed (Participants) | 22
years | 5.3 [3.0 to NA] — There have not been enough events occurring after the median was reached to estimate the upper limit of the confidence interval.

6. Secondary Outcome: Overall Survival (Cohort II)
Description: Estimated using the method of Kaplan-Meier.
Time Frame: Up to 10 years
Reporting Status: Not Posted

7. Secondary Outcome: Minimal Residual Disease Negativity
Description: To estimate in each cohort the rate of minimal residual disease (MRD) negativity.
Time Frame: as for outcome 4
Population: Only participants that had achieved CR or CRi and had available MRD data post-treatment were evaluated.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort I (Ph-) | Cohort II (Ph+/Ph-like)
Number analyzed (Participants) | 13 | 16
Participants
  MRD- | 12 | 7
  MRD+ | 1 | 9

8. Secondary Outcome: Time to Achieve Minimal Residual Disease Negativity
Description: Will be examined separately in descriptive analyses within each cohort.
Time Frame: Up to 10 years
Reporting Status: Not Posted

9. Secondary Outcome: Anti-idiotype Antibody Development
Description: To determine whether anti-idiotype antibodies directed against blinatumomab develop with blinatumomab treatment in this study.
Time Frame: Up to 10 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Duration of treatment and follow up until death or date of primary analysis (about 7.5 years)
Description: AEs and SAEs were reported using CTCAE v 4.0 and CTCAE v 5.0, respectively. The analysis populations for Adverse Events and All-Cause Mortality only differ for the Maintenance: Cohort I. The AE population includes participants that received maintenance treatment and thus does not include one participant which relapsed prior to receiving maintenance treatment. Whereas, the All-Cause Mortality population includes all participants registered to receive maintenance treatment.
Arm/Group | Induction: Cohort I (Ph-) | Induction: Cohort II (Ph+/Ph-like) | Post-remission: Cohort I (Ph-) | Post-remission: Cohort II (Ph+/Ph-like) | Maintenance: Cohort I (Ph-) | Maintenance: Cohort II (Ph+/Ph-like)
All-Cause Mortality (participants affected / at risk) | 1/29 | 2/24 | 0/19 | 0/18 | 0/14 | 1/16
Serious Adverse Events (participants affected / at risk) | 13/29 | 14/24 | 5/19 | 10/18 | 6/13 | 12/16
Other Adverse Events (participants affected / at risk) | 28/29 | 24/24 | 19/19 | 18/18 | 13/13 | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Induction: Cohort I (Ph-) (N=29) | Induction: Cohort II (Ph+/Ph-like) (N=24) | Post-remission: Cohort I (Ph-) (N=19) | Post-remission: Cohort II (Ph+/Ph-like) (N=18) | Maintenance: Cohort I (Ph-) (N=13) | Maintenance: Cohort II (Ph+/Ph-like) (N=16)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 1 | 3 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Chest pain - cardiac (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Heart failure (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 2
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 0
Eye disorders-Other (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 1 | 2
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Death NOS (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Edema limbs (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Fever (General disorders) | 1 | 3 | 2 | 1 | 3 | 0
General disorders and admin site conditions - Other (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Infusion related reaction (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cytokine release syndrome (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Catheter related infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0
Infections and infestations-Other (Infections and infestations) | 1 | 3 | 2 | 2 | 1 | 1
Lung infection (Infections and infestations) | 2 | 1 | 1 | 0 | 1 | 2
Sepsis (Infections and infestations) | 2 | 1 | 0 | 0 | 3 | 0
Upper respiratory infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Injury, poison and procedural complications - Other (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 2 | 0 | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 2 | 2 | 3 | 1
Platelet count decreased (Investigations) | 2 | 0 | 0 | 0 | 1 | 0
Weight loss (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
White blood cell decreased (Investigations) | 1 | 0 | 1 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Musculoskeletal and connective tiss disorder - Other (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nervous system disorders-Other (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Confusion (Psychiatric disorders) | 1 | 1 | 0 | 2 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 2 | 0 | 0 | 1 | 0
Hallucinations (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 | 0 | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 1 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 1 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 1 | 0
Hematoma (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 2
Hypotension (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0
Thromboembolic event (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Induction: Cohort I (Ph-) (N=29) | Induction: Cohort II (Ph+/Ph-like) (N=24) | Post-remission: Cohort I (Ph-) (N=19) | Post-remission: Cohort II (Ph+/Ph-like) (N=18) | Maintenance: Cohort I (Ph-) (N=13) | Maintenance: Cohort II (Ph+/Ph-like) (N=16)
Anemia (Blood and lymphatic system disorders) | 17 | 13 | 9 | 12 | 9 | 9
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 | 1 | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 6 | 1 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 3 | 2 | 2 | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 2 | 1 | 0 | 1 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cardiac disorders-Other (Cardiac disorders) | 1 | 1 | 0 | 1 | 2 | 1
Chest pain - cardiac (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Heart failure (Cardiac disorders) | 1 | 2 | 1 | 1 | 1 | 1
Palpitations (Cardiac disorders) | 0 | 2 | 0 | 2 | 2 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 2
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 2 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 4 | 2 | 4 | 3 | 3 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 2 | 0 | 0
Ear and labyrinth disorders-Other (Ear and labyrinth disorders) | 2 | 0 | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 2 | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 1
Endocrine disorders-Other (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 3
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 1 | 1 | 1 | 1 | 2
Blurred vision (Eye disorders) | 1 | 0 | 3 | 2 | 3 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 2
Dry eye (Eye disorders) | 2 | 0 | 2 | 0 | 1 | 1
Eye disorders-Other (Eye disorders) | 1 | 2 | 2 | 2 | 3 | 1
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Photophobia (Eye disorders) | 1 | 0 | 1 | 1 | 0 | 0
Retinopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Watering eyes (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 3 | 3 | 3 | 5 | 3
Anal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Bloating (Gastrointestinal disorders) | 4 | 1 | 1 | 1 | 1 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 10 | 4 | 2 | 4 | 8 | 4
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 5 | 8 | 2 | 9 | 5 | 11
Dry mouth (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 3 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Esophageal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Fecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 2
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 1
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 2 | 3 | 0 | 3 | 1 | 3
Hemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 6 | 1
Nausea (Gastrointestinal disorders) | 8 | 6 | 5 | 7 | 4 | 9
Oral hemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Rectal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Stomach pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 2
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2 | 2 | 4 | 3 | 4
Chills (General disorders) | 6 | 2 | 0 | 6 | 0 | 1
Edema face (General disorders) | 0 | 2 | 0 | 1 | 0 | 2
Edema limbs (General disorders) | 12 | 10 | 6 | 12 | 4 | 9
Edema trunk (General disorders) | 1 | 0 | 0 | 2 | 0 | 0
Fatigue (General disorders) | 12 | 13 | 5 | 12 | 8 | 9
Fever (General disorders) | 8 | 4 | 3 | 11 | 0 | 4
Flu like symptoms (General disorders) | 0 | 0 | 0 | 1 | 1 | 2
Gait disturbance (General disorders) | 0 | 0 | 0 | 2 | 0 | 2
General disorders and admin site conditions - Other (General disorders) | 3 | 1 | 1 | 5 | 2 | 3
Infusion related reaction (General disorders) | 1 | 0 | 0 | 0 | 1 | 0
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Irritability (General disorders) | 0 | 0 | 0 | 0 | 2 | 0
Localized edema (General disorders) | 0 | 1 | 0 | 2 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 2 | 0 | 1
Non-cardiac chest pain (General disorders) | 3 | 3 | 2 | 3 | 3 | 1
Pain (General disorders) | 1 | 4 | 4 | 3 | 2 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hepatobiliary disorders-Other (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Allergic reaction (Immune system disorders) | 0 | 1 | 0 | 1 | 0 | 1
Cytokine release syndrome (Immune system disorders) | 2 | 0 | 0 | 4 | 0 | 0
Immune system disorders-Other (Immune system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Conjunctivitis infective (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Infections and infestations-Other (Infections and infestations) | 1 | 0 | 0 | 1 | 5 | 1
Lung infection (Infections and infestations) | 1 | 2 | 1 | 0 | 2 | 1
Mucosal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Nail infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Skin infection (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0 | 2 | 0 | 2 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 1
Bruising (Injury, poisoning and procedural complications) | 3 | 3 | 0 | 1 | 3 | 0
Burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 2 | 2 | 2
Activated partial thromboplastin time prolonged (Investigations) | 3 | 1 | 2 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 10 | 5 | 4 | 4 | 7 | 2
Alkaline phosphatase increased (Investigations) | 4 | 5 | 3 | 3 | 3 | 4
Aspartate aminotransferase increased (Investigations) | 9 | 4 | 3 | 4 | 8 | 3
Blood bilirubin increased (Investigations) | 7 | 1 | 1 | 1 | 6 | 0
Cardiac troponin T increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0
Cholesterol high (Investigations) | 1 | 1 | 1 | 1 | 1 | 1
Creatinine increased (Investigations) | 6 | 4 | 2 | 3 | 3 | 4
Electrocardiogram QT corrected interval prolonged (Investigations) | 2 | 0 | 0 | 0 | 0 | 0
Fibrinogen decreased (Investigations) | 2 | 2 | 0 | 0 | 0 | 0
INR increased (Investigations) | 4 | 2 | 1 | 0 | 0 | 0
Investigations-Other (Investigations) | 3 | 2 | 4 | 3 | 1 | 4
Lymphocyte count decreased (Investigations) | 8 | 8 | 6 | 6 | 5 | 2
Lymphocyte count increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 5
Neutrophil count decreased (Investigations) | 13 | 14 | 6 | 9 | 11 | 4
Platelet count decreased (Investigations) | 15 | 16 | 7 | 3 | 10 | 1
Weight gain (Investigations) | 2 | 1 | 1 | 1 | 1 | 2
Weight loss (Investigations) | 1 | 1 | 3 | 1 | 0 | 2
White blood cell decreased (Investigations) | 15 | 12 | 7 | 9 | 7 | 2
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0
Anorexia (Metabolism and nutrition disorders) | 4 | 9 | 2 | 10 | 6 | 6
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 2 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 13 | 9 | 6 | 9 | 5 | 5
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 3 | 1 | 1 | 1 | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 1 | 0 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 1 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 13 | 13 | 7 | 7 | 8 | 6
Hypocalcemia (Metabolism and nutrition disorders) | 7 | 9 | 2 | 8 | 1 | 4
Hypoglycemia (Metabolism and nutrition disorders) | 4 | 1 | 3 | 0 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 6 | 5 | 1 | 3 | 3 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 5 | 3 | 3 | 2 | 2 | 0
Hyponatremia (Metabolism and nutrition disorders) | 13 | 3 | 4 | 1 | 3 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 3 | 8 | 1 | 6 | 1 | 1
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 3 | 7 | 3 | 4 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 0 | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 | 5 | 2 | 3 | 3 | 2
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1 | 0
Musculoskeletal and connective tiss disorder - Other (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 3 | 2 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 2 | 0 | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 1 | 2 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 2 | 2 | 3 | 6 | 4
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 2
Concentration impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 6 | 4 | 4 | 3 | 3 | 3
Dysarthria (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 2 | 3 | 1 | 0 | 0 | 1
Dysphasia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 7 | 8 | 8 | 7 | 5 | 6
Memory impairment (Nervous system disorders) | 0 | 0 | 3 | 1 | 3 | 2
Nervous system disorders-Other (Nervous system disorders) | 1 | 0 | 0 | 0 | 2 | 2
Paresthesia (Nervous system disorders) | 0 | 2 | 0 | 1 | 2 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 3 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 3 | 2 | 4 | 7 | 3
Sinus pain (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 2 | 5 | 1 | 1
Agitation (Psychiatric disorders) | 2 | 0 | 0 | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 5 | 3 | 2 | 2 | 1 | 2
Confusion (Psychiatric disorders) | 4 | 1 | 3 | 4 | 2 | 1
Delirium (Psychiatric disorders) | 3 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 3 | 0 | 2 | 0 | 3 | 1
Hallucinations (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 0
Insomnia (Psychiatric disorders) | 4 | 5 | 4 | 6 | 5 | 4
Acute kidney injury (Renal and urinary disorders) | 4 | 0 | 1 | 0 | 2 | 1
Chronic kidney disease (Renal and urinary disorders) | 1 | 1 | 1 | 0 | 0 | 0
Hematuria (Renal and urinary disorders) | 1 | 0 | 0 | 2 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Renal and urinary disorders-Other (Renal and urinary disorders) | 4 | 1 | 0 | 2 | 2 | 2
Renal calculi (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Urinary frequency (Renal and urinary disorders) | 5 | 2 | 1 | 2 | 2 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 1 | 1 | 1 | 1 | 1
Urinary retention (Renal and urinary disorders) | 0 | 2 | 0 | 1 | 0 | 1
Urinary urgency (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 1
Prostatic obstruction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 8 | 6 | 8 | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 | 12 | 3 | 9 | 7 | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 | 0 | 1 | 3 | 2 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 2 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 8 | 1 | 7 | 1 | 7
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 2 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 0 | 1 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Resp, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1 | 4 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 2 | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 1 | 4 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 2 | 1 | 3
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 0 | 1
Nail loss (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nail ridging (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 2 | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 2 | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 2 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 | 6 | 5 | 2 | 3 | 4
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2 | 1 | 3 | 4 | 3 | 3
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0
Surgical and medical procedures-Other (Surgical and medical procedures) | 0 | 0 | 0 | 2 | 0 | 3
Flushing (Vascular disorders) | 2 | 2 | 1 | 1 | 1 | 1
Hot flashes (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 0
Hypertension (Vascular disorders) | 8 | 2 | 5 | 5 | 4 | 4
Hypotension (Vascular disorders) | 4 | 2 | 0 | 3 | 3 | 0
Superficial thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Thromboembolic event (Vascular disorders) | 2 | 1 | 2 | 1 | 2 | 0
Vascular disorders-Other (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-16): https://cdn.clinicaltrials.gov/large-docs/14/NCT02143414/Prot_SAP_000.pdf